CLINICAL TRIAL: NCT03982953
Title: Predictors of Cognitive Change After Deep Brain Stimulation in the Subthalmic Nucleus in Parkinson's Disease
Brief Title: Predicting Cognition After DBS for Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dorothee Kübler, Postdoc and MD, Charite University, Berlin, Germany
Other Study IDs: EA2/040/19
Record Dates: First submitted 2019-06-09; First posted 2019-06-12 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Parkinson's Disease; Deep Brain Stimulation; Postoperativeneurocognitive Deficit; Postoperative Delirium
MeSH Terms: conditions — Parkinson Disease; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cholinergic biomarkers in cerebrospinal fluid (CSF)
  * TAU, phospho-TAU, ß-Amyloid 1-40 and 1-42
  * measured in CSF preoperatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD patients with STN-DBS: Patients with the diagnosis of Levodopa responsive idiopathic Parkinson's Disease that are planned to undergo craniectomy with implantation of bilateral DBS electrodes in the subthalamic nucleus
- Controls - PD patients with medical treatment: Patients with the diagnosis of Levodopa responsive idiopathic Parkinson's Disease that do not undergo DBS for personal reasons or contraindications for this treatment. Age, sex and disease-severity matched with PD patients with STN-DBS.

SUMMARY:
The aim of the study is to improve estimation of cognitive outcome after STN-DBS in PD in order to

* avoid risk factors by optimizing peri- and intraoperative management
* personalize therapeutic strategies for optimal long-term benefit

The investigators will test possible predictors (clinical, neuropsychological, neuroimaging, electrophysiological and molecular) for the risk of cognitive dysfunction after deep brain stimulation of the subthalamic nucleus (STN-DBS) in Parkinson's disease (PD) at a single center (Charité - Universitätsmedizin Berlin, Germany). Data collection takes place prior to as well as 3 and 12 months after the STN-DBS operation. Participation is proposed to all PD patients that are planned to undergo STN-DBS after careful examination of eligibility for this treatment according to standard operation procedures.

DETAILED DESCRIPTION:
Additionally to clinical routine tests, we will investigate the following possible predictors of cognitive dysfunction after STN-DBS in PD:

* Imaging biomarkers: volume of the nucleus basalis of Meynert (NBM) measured on preoperative MRI and data driven search for unknown MRI characteristics relating to the incidence of postoperative neurocognitive disorder by means of Deep Learning (Convolutional Neural Networks), test of previously established classification models
* Molecular biomarkers in CSF: TAU, phospho-TAU, ß-Amyloid 1-40 and 1-42 as well as NFL measured preoperatively
* Comorbidity: according to the Charlson Comorbidity Index
* Nutritional Status: defined by the Mini Nutritional Assessment (MNA-SF)
* Duration of intra-/perioperative brake of dopaminergic medication
* Nature and depth of anaesthesia: general or conscious sedation and depth of consciousness: as measured by 4 channel electroencephalography (SedLine®) and during implantation of impulse generator
* Incidence and duration of postoperative delirium: defined according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and/or as ≥ 2 points in the nursing Delirium Screening Scale (Nu-DESC) and/or a positive Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score, assessment three times daily during hospital stay
* Length of stay at ICU / hospital
* Postoperative organ complications: according to Clavien-Dindo classification
* Localisation of bilateral electrodes and active contacts on postoperative imaging

Substudies

Correlation of domain specific CANTAB connect test scores with possible predictors and incidence of postoperative neurocognitive disorder

Social Cognition: comparison of pre- and postoperative Theory of Mind (ToM) abilities measured by the Yoni-Paradigma (assesses affective and cognitive ToM)

The resulting multivariate risk model is expected

* to improve peri- and intraoperative management by identifying avoidable risk factors for the development of postoperative cognitive deficit
* to support evidence-based and personalized decision-making when advising PD patients considering STN-DBS
* to result in the development of future hypothesis-driven interventional trials on the basis of biomarker-based sub-grouping of patients
* to allow a better understanding of underlying pathophysiological processes both PD and surgery-related regarding cognitive effects of STN-DBS

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease
* Indication for STN-DBS

Exclusion Criteria:

* Internistic, surgical or psychiatric contrainidications with respect to the DBS operation or treatment for the STN-DBS group
* Dementia
* Relevant language barrier

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients that are planned to undergo STN-DBS. Possible contraindications to DBS are tested according to clinic-intern standard operation procedures. Tests include
  * Clinical scales: DemTect, MMST, ADL, MDS-UPDRS I-IV including video documentation of MDS-UPDRS III on and off dopaminergic medication
  * Questionnaires: expectations regarding DBS, PDQ39, BDI, Starkstein-Apathie-Skala, QUIP(-RS)
  * General examinations: Routine laboratory, ECG, TTE, Chest X-Ray, lung function, 24h-RR, Duplex sonography of extracranial arteries
  * Expert opinion from related fields: Neuropsychological exam, psychiatric examination, neurosurgery and anesthisiologic consultation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance after STN-DBS | Difference between pre- and 12 months postoperative testing
  Based on cognitive screening by paper pencil test (MoCA)
Incidence of postoperative neurocognitive disorder | Difference between pre- and 3 and 12 months postoperative testing
  • According to DSM-5 criteria applying the tablet-based neuropsychological test battery Cambridge Neuropsychological Test Automated Battery (CANTAB connect)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea A Kühn, Prof. MD, Study Director — Neurology, Head of the Movement Disorders and Neuromodulation Section
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kubler-Weller D, Stuke H, Astalosch M, Martins Ribeiro L, Landfried E, Schneider GH, Faust K, Krause P, Roediger J, Haufe S, Mousavi M, Al-Fatly B, Spies C, Borchers F, Kuhn AA. Predicting cognition after subthalamic Deep Brain Stimulation in Parkinson's Disease. NPJ Parkinsons Dis. 2025 Aug 28;11(1):265. doi: 10.1038/s41531-025-01128-3. PMID 40877314